CLINICAL TRIAL: NCT00059891
Title: Total Anorectal Reconstruction With The American Medical Systems, Inc. Acticon Neosphincter Prosthesis After Abdominoperineal Resection
Brief Title: Anal Sphincter Prosthesis in Treating Patients Who Are Undergoing Surgery for Anal or Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 02-124; P30CA008748 (NIH); MSKCC-02124
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Anal Cancer; Colorectal Cancer; Perioperative/Postoperative Complications
Keywords: perioperative/postoperative complications; stage II anal cancer; stage I anal cancer; stage III anal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Anus Neoplasms; Colorectal Neoplasms; Postoperative Complications; Rectal Neoplasms

ARMS (1):
- Anal Sphincter Prosthesis (Experimental): All patients will follow a common treatment algorithm. Anorectal reconstruction with the ABS neosphincter device will be a staged surgical approach. Routine postoperative testing will then be performed at 6 months (+/- 8 weeks) and 12 months (+/- 8 weeks), following ileostomy reversal which we have designated as time zero. Postoperative testing will include completion of a series of questionnaires.
  Interventions: Procedure: conventional surgery; Procedure: management of therapy complications

INTERVENTIONS:
Procedure: conventional surgery
Procedure: management of therapy complications

SUMMARY:
RATIONALE: An anal sphincter prosthesis may replace the need for a permanent colostomy and may improve the quality of life of patients who are undergoing surgery for anal or rectal cancer.

PURPOSE: Clinical trial to study the effectiveness of an anal sphincter prosthesis in treating patients who have anal or rectal cancer and are undergoing surgery to remove the anus and rectum.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the risk of complications and feasibility of total anorectal reconstruction using the Acticon Neosphincter prosthesis after abdominoperineal resection in patients with anal or rectal cancer.
* Determine continence, bowel function, and quality of life of patients treated with this surgery.

OUTLINE: Patients undergo abdominoperineal resection (APR) with perineal colostomy and diverting loop ileostomy. At least 3 months after APR, patients undergo placement of the Acticon Neosphincter prosthesis. At least 6 weeks after prosthesis placement, the prosthesis is activated. When the patient demonstrates the ability to operate the prosthesis, the ileostomy is reversed.

Quality of life is assessed at 6 and 12 months and then annually thereafter.

Patients are followed at 6 and 12 months and then annually thereafter.

ELIGIBILITY:
Subject Inclusion Criteria:

* Histologically proven cancer of distal rectum or anus
* Not candidates for sphincter preservation
* > or = 18 years of age
* an acceptable risk for surgery and general anesthesia
* sufficient dexterity and mental capacity to operate the device
* willing and able to give valid Informed Consent

Subject Exclusion Criteria:

* Patients with recurrent anorectal cancer
* Patients with metastatic anorectal cancer
* Patients at high risk for local recurrence
* Patients with active pelvic sepsis
* Patients currently enrolled in another study involving an investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Determine the risk of complications and feasibility of total anorectal reconstruction using the Acticon Neosphincter prosthesis after abdominoperineal resection in patients with anal or rectal cancer. | 2 years

SECONDARY OUTCOMES:
Determine continence, bowel function, and quality of life of patients treated with this surgery. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: W. Douglas Wong, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States